CLINICAL TRIAL: NCT04996628
Title: Pancreatic Quantitative Sensory Testing (P-QST) to Predict Treatment Response for Pain in Chronic Pancreatitis
Acronym: P-QST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Anna Evans Phillips, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY21050169; R01DK127042 (NIH)
Record Dates: First submitted 2021-07-23; First posted 2021-08-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pancreatitis; Chronic Pain
Keywords: Chronic Pain; Chronic Pancreatitis; Recurrent Acute Pancreatitis; Chronic Abdominal Pain; ERCP; Pancreatic Surgery
MeSH Terms: conditions — Pancreatitis, Chronic; Chronic Pain; Pancreatitis | interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Intervention Model Description: Participants are assessed at baseline for nociceptive pattern via P-QST and followed longitudinally for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pancreatic Quantitative Sensory Testing (P-QST) (Experimental): Definite Chronic Pancreatitis patients undergoing decompressive invasive treatments (endoscopic therapy or surgery) to relieve main pancreatic duct obstruction due to stones and/or stricture for management of pain will undergo P-QST prior to clinically-indicated invasive treatment.
  Interventions: Diagnostic Test: Quantitative Sensory Test 1; Diagnostic Test: Quantitative Sensory Test 2; Diagnostic Test: Quantitative Sensory Test 3

INTERVENTIONS:
Diagnostic Test: Quantitative Sensory Test 1 — Subject will give pain rating (on Visual Analogue Scale (VAS) 0-10) of single as well as multiple stimulation with round-tip non-invasive pin-prick device. Difference is recorded as Temporal Summation Score.
  Other Names: Temporal Summation
Diagnostic Test: Quantitative Sensory Test 2 — Subject will state when they first detect pain and pain detection threshold in response to pressure administration with pressure algometer. Pressure threshold recorded in kilopascals(kP). Stimulation will be repeated in pancreatic and control dermatomes. Subject will then state pain tolerance threshold at same locations. Sensitization will be characterized by ratio of pancreatic vs. control dermatome scores.
  Other Names: Pressure Threshold Testing
Diagnostic Test: Quantitative Sensory Test 3 — Subject will apply dominant hand to ice-chilled water bath (36F) for up to 2 minutes. Pain score (VAS 0-10) will be assessed each 10 seconds. Pain tolerance threshold (in kP) will be assessed with algometer on non-dominant thigh before and after water bath to determine change in threshold. Difference in pain tolerance recorded as Conditioned Pain Modulation Score.
  Other Names: Conditioned Pain Modulation

SUMMARY:
Abdominal pain in chronic pancreatitis (CP) affects up to 90% of patients during the course of their disease, and response to currently available therapies is suboptimal and unpredictable. The proposed clinical trial will evaluate the predictive capability of Pancreatic Quantitative Sensory Testing (P-QST) - a novel assessment of neurosensory phenotyping- for improvement in pain in patients with CP who are undergoing medically-indicated invasive treatment with endoscopic therapy or surgery.

DETAILED DESCRIPTION:
P-QST has been shown to be able to phenotype patients with CP into nociceptive patterns according to degree of central sensitization. As a tool to identify baseline nociceptive pattern in patients with painful CP, P-QST will be performed at baseline prior to planned invasive treatment with endoscopic therapy or decompressive surgery. We will evaluate the ability of P-QST to predict response to invasive treatment for painful CP, and to develop a predictive model for individualized prediction of treatment response.

Patients will undergo pre-procedure P-QST testing before undergoing scheduled invasive treatment as directed by their treating gastroenterologist. The date of first endoscopic therapy or surgery will be used to calculate follow-up timepoints, which will be scheduled at 3, 6, and 12 months after the first endotherapy session or surgery. At each follow-up time point, patients will answer questions about their pain. In addition, patients will complete patient reported outcome tools (HADS, PCS instruments) and the Patient Global Impression of Change. Serum and urine samples will be obtained at baseline and at 6-month follow-up timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age with definite CP undergoing decompressive invasive treatments (endoscopic therapy or surgery) to relieve main pancreatic duct obstruction due to stones and/or stricture for management of pain.

  * Endoscopic therapy: Endoscopic Retrograde Cholangiopancreatography (ERCP) with pancreatic duct stone removal, stent placement, and/or stricture dilation, ± intraductal lithotripsy or Extracorporeal Shock Wave Lithotripsy (ESWL).
  * Surgery: drainage procedures (Frey and Puestow operations)

Exclusion Criteria:

* Patients with chronic pain from conditions other than CP
* Patients < 18 years of age
* Patients who have had endoscopic therapy within the past 12 months
* Patients who have undergone prior pancreatic surgery
* Patients who have resective surgical procedure planned (eg. Whipple procedure, Total Pancreatectomy)
* Patients with peripheral sensory deficits
* Patients with known pregnancy at the time of study screening**

  * Note: Women who become pregnant during the course of the study can no longer participate in P-QST testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Average Pain Score | six months post procedure
  The primary outcome of the study is average pain score at 6 months post-procedure based on single-question numeric rating scale (NRS) (Scale of 0 to 10 how intense abdominal pain has been on average over the past 7 days (Scale: 0=No pain, 10=Worst pain Imaginable.)

SECONDARY OUTCOMES:
Change from baseline in Seven Day Pain Diary Score | 3 months after intervention.
  The 7-day pain diary average score at 3 months after intervention. (Scale 0 = no pain to 10 = worst pain imaginable)
Change from baseline in Seven Day Pain Diary Score | 6 months after intervention.
  The 7-day pain diary average score at 6 months after intervention. (Scale 0 = no pain to 10 = worst pain imaginable)
Change from baseline in Seven Day Pain Diary Score | 12 months after intervention.
  The 7-day pain diary average score at 12 months after intervention. (Scale 0 = no pain to 10 = worst pain imaginable)
Change from baseline in Single-question NRS score | at 3 months after intervention
  Single-question NRS at 3 months after intervention (Scale 0 = no pain to 10 = worst pain imaginable)
Change from baseline in Single-question NRS score | at 12 months.
  Single-question NRS at 12 months after intervention (Scale 0 = no pain to 10 = worst pain imaginable)
Number of patients using prescription opioids for pain control at time of assessment | 3 months
  Opioid use (yes,no binary answer) at 3 months.
Number of patients using prescription opioids for pain control at time of assessment | 6 months
  Opioid use (yes,no) at 6 months.
Number of patients using prescription opioids for pain control at time of assessment | 12 months
  Opioid use (yes,no) at 12 months.
Mean reported daily opioid dose for patients using prescription opioids at time of assessment | 3 months
  Opioid dose (continuous variable in milligrams of morphine equivalent) at 3 months.
Mean reported daily opioid dose for patients using prescription opioids at time of assessment | 6 months
  Opioid dose (continuous variable in milligrams of morphine equivalent) at 6 months.
Mean reported daily opioid dose for patients using prescription opioids at time of assessment | 12 months
  Opioid dose (continuous variable in milligrams of morphine equivalent) at 12 months.
Pain relief of ≥30% | 3 months
  Percentage of patients with ≥30% at 3 months after intervention
Pain relief of ≥30% | 6 months
  Percentage of patients with ≥30% at 6 months after intervention
Pain relief of ≥30% | 12 months
  Percentage of patients with ≥30% at 12 months after intervention
Pain relief of ≥50% | 3 months after intervention
  Percentage of patients with ≥50% at 3 months after intervention.
Pain relief of ≥50% | 6 months after intervention
  Percentage of patients with ≥50% at 6 months after intervention.
Pain relief of ≥50% | 12 months after intervention
  Percentage of patients with ≥50% at 12 months after intervention.
Change from baseline on the Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale | Baseline, 3, 6, and 12 months
  The PROMIS Global Health Questionnaire is a validated self-reported tool that scores both mental and physical health at the time of assessment. Possible scores for both Mental and Physical Health range from 7 to 35 (lower score corresponds to poorer physical or mental health).
Change from baseline on the Patient Reported Outcomes Measurement Information System (PROMIS) Neuropathic Pain Scale | Baseline, 3, 6, and 12 months
  The PROMIS Global Health Questionnaire is a validated self-reported tool that scores neuropathic pain characteristics at the time of assessment. Possible scores range from 5 to 25 (higher score corresponds to more neuropathic pain characteristics).
Change from baseline on the Patient Reported Outcomes Measurement Information System (PROMIS) Nociceptive Pain Scale | Baseline, 3, 6, and 12 months
  The PROMIS Global Health Questionnaire is a validated self-reported tool that scores nociceptive pain characteristics at the time of assessment. Possible scores range from 5 to 25 (higher score corresponds to more nociceptive pain characteristics).
Change from baseline on the Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Scale | Baseline, 3, 6, and 12 months
  The PROMIS Global Health Questionnaire is a validated self-reported tool that scores pain interference with aspects of daily life at the time of assessment. Possible scores range from 6 to 30 (higher score corresponds to more pain interference with daily activities).
Patient Global Impression of Change (PGIC) Scale | 3, 6, and 12 months
  The PGIC is a validated self-reported tool that scores the patient's impression of change from baseline of their pain and overall health. Possible scores range from 1 to 7 (higher score corresponds to improvement).
Change from baseline on the Pain Catastrophizing Scale (PCS) | Baseline, 3, 6, and 12 months
  The PCS is a validated self-reported tool that scores the patient tendency to catastrophize about pain or potential pain. Possible scores range from 0 to 42 (higher scores reflect more catastrophizing tendencies).
Change from baseline on the Hospital Anxiety and Depression Scale (HADS) | Baseline, 3, 6, and 12 months
  The HADS is a validated self-reported tool that screens for symptoms of anxiety and depression. Possible scores range from 0 to 21 (higher scores reflect more severe symptoms of anxiety or depression).
Change from baseline on the Modified Brief Pain Inventory Short Form (mBPI-SF) | Baseline, 3, 6, and 12 months
  The mBPI-SF is a validated self-reported tool that evaluates pain severity and pain interference with daily activities at the time of assessment. Possible scores for pain severity range from 0 to 40 (higher scores reflect more severe pain); possible scores for pain interference range from 0 to 70 (higher scores reflect more pain interference with daily life).
Change from baseline on the European Organization for the Research and Treatment of Cancer Quality(EORTC) of Life Questionnaire (QLQ) Core 30 (C30) | Baseline, 3, 6, and 12 months
  The EORTC QLQ-C30 is a validated self-reported tool measuring quality of life that reports scores on global health (quality of life), functioning (physical, role, emotional, cognitive, social), and symptoms (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). All scores range from 0 to 100. A high score on quality of life indicates higher quality of life; a high score on a functioning scale indicates a higher level of functioning, and a high score on a symptom scale indicates a higher level of symptoms.
Change from baseline on the Comprehensive Pain Assessment Tool for Pancreatitis Short Form (COMPAT-SF) | Baseline, 3, 6, and 12 months
  The COMPAT-SF is a validated self-reported tool specifically designed for patients with pancreatic disease. Scores for pain severity (average, worst, and least) range from 0 to 10 (higher corresponds to more pain); scores for pain triggers (including food, exercise, and thermal changes) are scored on a scale from never to always (never, rarely, sometimes, very often, always); scores for pain symptom characteristics (cramping, shooting, stabbing) are scored on a scale from 0 (none) to 10 (worst possible).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Evans Phillips, MD, MS, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Indiana University Medical Center, Indianapolis, Indiana
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data may be shared with investigators from outside institutions for ancillary studies upon request. Requests should be made to study principal investigator at evansac3@upmc.edu.
  Researchers interested in learning techniques of P-QST will be able to receive information and training upon request through our institutions. Results and conclusions from this project will be shared publicly with other medical research and physicians through presentation at scientific meetings and in one or more final publications.
Time Frame: Data will be available at the close of the study and for 5 years subsequent.
Access Criteria: Individual requests for data sharing can be made to evansac3@upmc.edu

REFERENCES:
- [Derived] Phillips AE, Afghani E, Akshintala VS, Benos PY, Das R, Drewes AM, Easler J, Faghih M, Gabbert C, Halappa V, Khashab MA, Olesen SS, Saloman JL, Sholosh B, Slivka A, Wang T, Yadav D, Singh VK. Pancreatic quantitative sensory testing to predict treatment response of endoscopic therapy or surgery for painful chronic pancreatitis with pancreatic duct obstruction: study protocol for an observational clinical trial. BMJ Open. 2024 Mar 21;14(3):e081505. doi: 10.1136/bmjopen-2023-081505. PMID 38514147